CLINICAL TRIAL: NCT03707054
Title: Correlation Between Vasopressin and Renal Function Following a Controlled Intraabdominal Pressure Elevation
Brief Title: Vasopressin in Intraabdominal Pressure Elevation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Emanuele LoMenzo, Principal Investigator, The Cleveland Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: FLA 17-031
Record Dates: First submitted 2018-06-22; First posted 2018-10-16 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Intracranial Pressure Increase; Abdominal Compartment Syndrome
MeSH Terms: conditions — Intracranial Hypertension; Intra-Abdominal Hypertension

STUDY DESIGN:
Intervention Model Description: prospective trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Study Arm (Experimental): Measurements of optic nerve diameter, Urine and plasma osmolality, Serum vasopressin.
  Interventions: Diagnostic Test: Study Arm

INTERVENTIONS:
Diagnostic Test: Study Arm — Measurements of optic nerve diameter, serum and urine osmolarity, serum vasopressin

SUMMARY:
The aim of this study is to investigate any direct correlation between increased intrathoracic pressure, intraabdominal pressure and intracranial pressure, following a controlled elevation in intraabdominal pressure and intrathoracic pressure (PEEP). The second end-point is to investigate any correlation between elevated intracranial pressure and vasopressin release, urine output and urine and serum osmolality by measuring their values at different time-points.

DETAILED DESCRIPTION:
Increase in intraabdominal pressure (IAP) has been demonstrated to correlate with consequential hemodynamic effects. Several studies have been carried out mostly in experimental settings to define the underlying mechanisms that regulate the pathophysiology following an increase in IAP. In the last years this topic has become concerning because of the wide spread of laparoscopy, that is namely an iatrogenic acute increase in IAP.

Patients selected and consented for elective surgery will undergo standard of care and additional measurements during and after surgery. The measurements will be done at different stages of laparoscopic surgery.

1. A) Baseline, patient under general anesthesia, Foley catheter positioned, beginning urine collection, before insufflation of pneumoperitoneum
2. B) 10-15 minutes after insufflation of pneumoperitoneum at 15mmHg, PEEP at 5cmH2O or lowest setting
3. C) 10-15 minutes after stabilization of PEEP at 10cmH2O, pneumoperitoneum still at 15 mmHg
4. D) 10-15 minutes after desufflation of pneumoperitoneum and basal mechanical ventilation

Measurements include :

* Intraabdominal pressure IAP: assessed via laparoscopic insufflator, set at 15 mmHg as a standard value for all laparoscopic procedures
* Intrathoracic pressure: indirectly measured by variability of peak expiratory pressures
* Urine collection: through a Foley catheter from the beginning of surgery to post-operative day 1
* Urine osmolality (to be assessed at set time-points )
* Hourly urine output (at least 24 hours in order to evaluate expected significant variation even after the procedure end, since renal adaptation could take longer period)
* Serum/plasma collection : blood draws to evaluate specific values of
* Plasma Vasopressin (ADH)
* Serum osmolality
* Mean arterial pressure : standard of care
* Pulmonary expiratory end-pressure (PEEP): anesthesiologists routinely adapt PEEP in order to maintain an optimal ventilation, especially in obese patients and during laparoscopy
* Optic nerve sheath diameter (ONSD): a 7.5-MHz linear ultrasound probe to measure the diameter of the optic nerve sheath 3 mm behind the globe is going to be used; a trained study personnel physician will take the non-invasive sonographic picture using ultrasound. The ONSD will be measured from the captured picture. Study personnel will record the interaction on the patient's chart and include the measurement on the database

ELIGIBILITY:
Inclusion Criteria:

* Age 18-72
* Patients meeting NIH criteria for bariatric surgery
* Patients undergoing laparoscopic sleeve gastrectomy

Exclusion Criteria:

* • Age below 18 years

  * American Society of Anesthesiologist (ASA) class IV or V
  * Other evident/diagnosed causes of increased IAP or increased intrathoracic pressure, except for obesity
  * Active urinary tract infection
  * Previous or concomitant neurological disease
  * Previous or concomitant ophthalmic conditions/eye surgery
  * Previous or concomitant lung diseases

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-04-28 (Actual); Primary Completion 2024-05-28 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Physiologic variations secondary to pneumoperitoneum | 24 hours
  The investigators will measure the intrabdominal pressure (IAP) pressure using the laparoscopic insufflator dial, the optic nerve sheath diameter (OSND) using an ultrasound which is a surrogate of the intracranial pressure (ICP), the variation of vasopressin levels, and the urine osmolality at baseline and during pneumoperitoneum. This is done in an effort to understand the compensatory measure used during pneumoperitoneum and abdominal compartment syndrome

CONTACTS AND LOCATIONS:
Locations (1):
- Cleveland Clinic Florida, Weston, Florida, United States

IPD SHARING:
Plan to Share IPD: No